CLINICAL TRIAL: NCT07227584
Title: Treatment of Newly Diagnosed Philadelphia Chromosome-Negative Acute Lymphoblastic Leukemia in Adolescents and Young Adults (AYAs)
Brief Title: ALL Backbone in AYAs
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Marlise Luskin, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25-533
Record Dates: First submitted 2025-11-10; First posted 2025-11-12 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Acute Lymphoblastic Leukemia; Philadelphia Chromosome-Negative Lymphoblastic Leukemia; Acute Lymphoblastic Leukemia (ALL); Leukemia
Keywords: Acute Lymphoblastic Leukemia; Philadelphia Chromosome-Negative lymphoblastic leukemia; Acute Lymphoblastic Leukemia (ALL); Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia | interventions — blinatumomab; pegaspargase; Cyclophosphamide; Cytarabine; Dexamethasone; Calcium Dobesilate; Doxorubicin; Etoposide; etoposide phosphate; Mercaptopurine; Methotrexate; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ALL Backbone Regimen for B-Cell (Experimental): * Steroid Prophase (3-dy cycle): Dexamethasone & cytarabine
  * Induction IA (29-dy cycle): Vincristine, dexamethasone, pegaspargase, doxorubicin, IT chemotherapy
  * Induction IB (42-dy cycle): Cyclophosphamide, cytarabine, mercaptopurine, IT chemotherapy
  * Blinatumomab Cycle 1, 2 (42-dy cycles): Blinatumomab, dexamethasone, IT chemotherapy
  * Consolidation I:
    * Phase IA (28-dy cycle), Phase IC (21-dy cycle): Vincristine, mercaptopurine, methotrexate, dexamethasone, cytarabine, etoposide, pegaspargase, IT chemotherapy
  * Blinatumomab Cycle 3 (42-dy cycle): Dexamethasone, Blinatumomab, IT chemotherapy
  * Consolidation II (21-dy cycles for 30 wks): Vincristine, dexamethasone, mercaptopurine, doxorubicin, methotrexate, pegaspargase, IT chemotherapy
  * Blinatumomab Cycle 4 (42-dy cycle): Dexamethasone, Blinatumomab, IT chemotherapy
  * Continuation (21-dy cycles): Vincristine, dexamethasone, mercaptopurine, methotrexate, IT chemotherapy
  * End of treatment visit
  * Follow up
  Interventions: Drug: Blinatumomab; Drug: Oncaspar; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dexamethasone; Drug: Doxorubicin Hydrochloride; Drug: Etoposide; Drug: Mercaptopurine; Drug: Methotrexate
- ALL Backbone Regimen for T-Cell (Experimental): * Steroid Prophase (3-day cycle): Dexamethasone and cytarabine
  * Induction IA (29-day cycle): Vincristine, dexamethasone, pegaspargase, doxorubicin, IT chemotherapy
  * Induction IB (42-day cycle): Cyclophosphamide, cytarabine, mercaptopurine, IT chemotherapy
  * Consolidation I:
    * Phase IA (28-day cycle) and Phase IC (21-day cycle): Vincristine, mercaptopurine, methotrexate, dexamethasone, cytarabine, etoposide, pegaspargase, IT chemotherapy
  * CNS Phase (21-day cycle): Dexamethasone, vincristine, mercaptopurine, pegaspargase, IT chemotherapy
  * Consolidation II (21-day cycles for 30 weeks): Vincristine, dexamethasone, mercaptopurine, doxorubicin, methotrexate, pegaspargase, IT chemotherapy
  * Continuation (21-day cycles): Vincristine, dexamethasone, mercaptopurine, methotrexate, IT chemotherapy
  * End of treatment visit
  * Follow up
  Interventions: Drug: Blinatumomab; Drug: Oncaspar; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dexamethasone; Drug: Doxorubicin Hydrochloride; Drug: Etoposide; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Vincristine

INTERVENTIONS:
Drug: Blinatumomab — A bispecific T-cell engager (BiTE) antibody, single-use vial via intravenous infusion, per standard of care
  Other Names: Blincyto; NSC# 765986
Drug: Oncaspar — A modified enzyme L-asparaginase, single-use vial via intravenous infusion, per standard of care
  Other Names: PEGASPARGASE; NSC #624239)
Drug: Cyclophosphamide — An alkylating agent, single-use vial via intravenous infusion, per standard of care
  Other Names: Cytoxan; NSC #26271
Drug: Cytarabine — An antineoplastic antimetabolite, multi-dose vial via intrathecal injection (through the spinal space), per standard of care
  Other Names: Cytosine Arabinoside; Ara-C; Cytostar; NSC#63878
Drug: Dexamethasone — A synthetic glucocorticoid, tablets or single-use vials via orally or intravenous infusion (through the vein), per standard of care
  Other Names: Decadron; Hexadrol; Dexone; Dexameth; NSC#34521
Drug: Doxorubicin Hydrochloride — An anthracycline antibiotic, single-use or multi-dose vials via intravenous infusion, per standard of care
  Other Names: Adriamycin; NSC#123127
Drug: Etoposide — A derivative of podophyllotoxin, multi-dose vial via intravenous infusion, per standard of care
  Other Names: VePesid; Etopophos; VP-16; NSC#141540
Drug: Mercaptopurine — A purine antagonist, tablet via orally, per standard of care
  Other Names: 6-MP; Purinethol; 6-Mercaptopurine; Purixan; NSC#000755
Drug: Methotrexate — A folate analogue, multi-dose and single-use vials via intrathecal injection, per standard of care
  Other Names: MTX; Amethopterin; Trexall; NSC#000740
Drug: Vincristine — A vinca alkaloid, single-use vials via intravenous injection, per standard of care
  Other Names: Oncovin; VCR; LCR; NSC#67574
  Arms: ALL Backbone Regimen for T-Cell

SUMMARY:
The goal of this research study is to evaluate a chemotherapy regiment for the treatment of newly diagnosed Philadelphia chromosome-negative acute lymphoblastic leukemia (ALL) in adolescents and young adults (AYAs).

The names of the study drugs involved in this study are:

* blinatumomab (a type of immunotherapy drug)
* cyclophosphamide (a type of chemotherapy drug)
* cytarabine (a type of antineoplastic agent)
* dexamethasone (a type of synthetic glucocorticoid)
* doxorubicin (a type of antineoplastic agent)
* etoposide (a type of antineoplastic agent)
* mercaptopurine (a type of antineoplastic agent)
* methotrexate (a type of chemotherapy drug)
* pegaspargase (a type of antineoplastic agent)
* vincristine (a type of antineoplastic agent)

DETAILED DESCRIPTION:
This Phase 2, single-arm research study is to evaluate a chemotherapy regiment the treatment of newly diagnosed Philadelphia chromosome-negative acute lymphoblastic leukemia (ALL) in adolescents and young adults (AYAs).

The U.S. Food and Drug Administration (FDA) has approved all of the drugs of treatment being studied but the investigators of this research study want to understand more about the safety and effectiveness of the chemotherapy regimen in adolescents and young adults with newly diagnosed Philadelphia chromosome-negative ALL.

The research study procedures include screening for eligibility, in-clinic visits, blood tests, urine tests, saliva tests, X-rays, electrocardiograms (ECGs), echocardiograms (ECHOs), Dual-Energy X-ray Absorptiometry (DEXA) scans, bone marrow aspirations/biopsies.

Participation in this study is expected to last about 10 years, 2 years of treatment followed by 8 years of follow up.

It is expected that about 67 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

3.1.1Confirmed diagnosis of Philadelphia chromosome-negative acute lymphoblastic leukemia.

* Diagnosis should be made by peripheral blood, bone marrow aspirate, bone marrow biopsy, or tissue biopsy demonstrating ≥25% involvement by lymphoblasts, with flow cytometry or immunohistochemistry confirming B-ALL or T-ALL.

  o Participants with B-cell and T-cell lymphoblastic lymphoma are eligible regardless of bone marrow involvement Participants with mixed phenotype acute leukemia (MPAL) ARE eligible, if an ALL regimen is felt to be most appropriate treatment.
* Participants with CNS leukemia ARE eligible. 3.1.2 Allowed prior therapy:
* Corticosteroids, hydroxyurea, all-trans retinoic acid (ATRA).
* IT chemotherapy.
* Emergent radiation therapy or leukapheresis for life threatening complications.
* One cycle of prior chemotherapy (i.e. an induction cycle given at another institution and participant transfers care for post-induction treatment; OR a participant does not meet eligibility prior to induction but does meet eligibility after remission induction).

3.1.3 Age 18.00 - 50.99 years 3.1.4 Direct bilirubin <1.4 mg/dL (total bilirubin < 1.4 mg/dL is acceptable). 3.1.5 Willingness to use effective means of birth control. The effects of chemotherapy on the developing human fetus are unknown. For this reason and because therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of study.

3.1.6 Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

Philadelphia chromosome-positive / BCR::ABL1 fusion 3.2.2 Participants with mature B-cell (Burkitt's) ALL. Mature B-cell ALL is defined by the presence of surface immunoglobulin AND any of the following: t(8;14)(q24;q32), t(8;22), t(2;8), or c-myc-gene rearrangement by FISH, PCR or other testing. [FISH/PCR testing for c-myc rearrangements is not required prior to study entry, but it is suggested for participants with surface immunoglobulin expression or L3 morphology]. 3.2.3 Participants with acute undifferentiated leukemia. 3.2.4 Participants receiving any other investigational agent for this condition.

3.2.5 Uncontrolled intercurrent illness including but not limited to ongoing infection with vital sign instability (hypotension, respiratory insufficiency), life-threatening acute tumor lysis syndrome (e.g., with renal failure), symptomatic congestive heart failure, cardiac arrhythmia, intracranial or other uncontrolled bleeding. Circumstances that may significantly interfere with a participant's ability to safely comply with study procedures, such as attend scheduled study visits, adhere to treatment protocols, or complete study assessments. These include a lack of reliable transportation, unstable housing, or psychiatric illness, but reasonable attempts should be made to overcome these circumstances, including but not limited to identifying sponsor, institutional, or thirdparty financial or social support as well as psychiatric consultation for objective assessment. 3.2.6 Sexually active participants of reproductive potential who have not agreed to use an effective contraceptive method for the duration of study participation are ineligible.

3.2.7 Pregnant women are excluded from this study because many of the agents used on this protocol have potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with these chemotherapy agents, breastfeeding should be discontinued if the mother is enrolled.

Ages: 18 Years to 51 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 67 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2030-07-31 (Estimated); Study Completion 2035-07-31 (Estimated)

PRIMARY OUTCOMES:
Treatment Completion Rate Through Time Point 3 (TP3) | Timeframe for TP3 depends on disease immunophenotype. Participants with CD19-positive B-ALL, TP3 occurs at the end of Blinatumomab Cycle 2 on Day 28 (130 days from study start). For participants with T-cell ALL or those who do not receive blinatum
  Treatment completion rate through TP3 is defined as the proportion of Adolescents and Young Adults (AYAs) participants who receive all protocol-specified therapy through TP3, without early discontinuation.

SECONDARY OUTCOMES:
Rate of Treatment-Related Mortality (TRM) | Up to 115 weeks
  Rate of TRM is defined as the proportion of participants who die due to treatment-related causes.
Rate of Treatment Discontinuation due to Toxicity or Disease | Up to 115 weeks
  Rate of treatment discontinuation during Induction, Consolidation, and Continuation phases, defined as the proportion of participants who stop protocol-specified therapy due to regimen-related toxicity and/or treatment failure.
Rate of Asparaginase Non-Completion | This endpoint is assessed during Consolidation II, which occurs approximately from Day 270 to Day 480 of study treatment.
  Rate of asparaginase non-completion is defined as the proportion of participants who did not complete all planned doses of asparaginase per protocol.
Reason of Asparaginase Non-Completion | Up to 115 weeks
  This outcome summarizes the reasons participants discontinue asparaginase treatment earlier than planned.
Grade 3 Infections Toxicity Rate | Adverse events will be followed for 30 days after completion of protocol treatment, with the overall treatment period up to 115 weeks.
  Grade 3 infection toxicity rate is defined as the proportion of participants who experience grade 3 bacterial or fungal infections that are assessed as possibly, probably, or definitely related to the study treatment during the induction, consolidation, and continuation phases. Toxicity grades are determined according to the Common Terminology Criteria for Adverse Events (CTCAE) version 6.0.
Grade 3 Asparaginase-associated Toxicities Rate | Adverse events will be followed for 30 days after completion of protocol treatment, with the overall treatment period up to 115 weeks.
  Grade 3 asparaginase-associated toxicity rate is defined as the proportion of participants who experience grade 3 asparaginase-associated toxicities (including thromboembolic events, pancreatitis, hypertriglyceridemia, hyperbilirubinemia, hypersensitivity, and hyperglycemia) that are assessed as possibly, probably, or definitely related to the study treatment during the induction, consolidation, or continuation phases. Toxicity grades are determined according to the Common Terminology Criteria for Adverse Events (CTCAE) version 6.0.
Grade 3 Orthopedic Toxicity Rate | Adverse events will be followed for 30 days after completion of protocol treatment, with the overall treatment period up to 115 weeks. Ostenonecrosis and fractures will be followed up to 10 years.
  Grade 3 orthopedic toxicity rate is defined as the proportion of participants who experience grade 3 osteopenia or osteoporosis that are assessed as possibly, probably, or definitely related to the study treatment at the end of treatment, or osteonecrosis (ON) or fractures during or after treatment. Toxicity grades are assigned according to the Common Terminology Criteria for Adverse Events (CTCAE) version 6.0.
Complete remission Rate (CRR) | CR can be documented either at the end of Induction IA (32 days) or Induction IB (74 days).
  CRR is defined as proportion of participants who achieve CR. Complete response (CR) is defined as an interpretable bone marrow with less than 5% malignant lymphoblasts, no lymphoblasts in peripheral blood, an absolute phagocyte count greater than 1000/µL and platelets above 100,000/µL (for participants with M2 marrow at Day 32 who achieve CR at TP2, APC above 500/µL and platelets above 50,000/µL are acceptable), no evidence of extramedullary leukemia or blasts in spinal fluid, at least a 70% reduction in the anterior mediastinal mass if present at diagnosis as measured by the sum of the products of the two greatest diameters on CT or chest X-ray, and for any other large radiographic masses at diagnosis, a 70% reduction in SPD if restaging imaging is obtained.
Measurable Residual Disease (MRD) Negativity Rate at the end of Induction IA (Time Point 1) | At the end of Induction IA (32 days from study start)
  The proportion of who achieve measurable residual disease (MRD) negativity at the end of Induction IA (Time Point 1). MRD negativity is assessed by multiparameter flow cytometry (MPFC), next-generation sequencing (NGS), and/or KMT2A::AFF4 RT-PCR.
Measurable Residual Disease (MRD) Negativity Rate at the end of Induction IB (Time Point 2) | At the end of Induction IB (74 days from study start)
  The proportion of who achieve measurable residual disease (MRD) negativity at the end of Induction IB (Time Point 2). MRD negativity is assessed by multiparameter flow cytometry (MPFC), next-generation sequencing (NGS), and/or KMT2A::AFF4 RT-PCR.
Measurable Residual Disease (MRD) Negativity Rate at Time Point 3 (TP3) | For CD19-positive B-ALL, TP3 is reached at the end of Blinatumomab Cycle 2 on Day 28 (Day 130 from study start). For T-cell ALL or participants not receiving blinatumomab, TP3 occurs on Day 28 of Consolidation IC (Day 102 from study start).
  The proportion of who achieve measurable residual disease (MRD) negativity at TP3. MRD negativity is assessed by multiparameter flow cytometry (MPFC), next-generation sequencing (NGS), and/or KMT2A::AFF4 RT-PCR.
Median Event-Free Survival (EFS) | Up to 10 years
  EFS based on Kaplan-Meier method is defined as the time from registration to induction failure, relapse, second malignancy, or death due to any cause. Relapse is defined as the presence of more than 5% lymphoblasts in bone marrow confirmed by flow cytometry, cytogenetics, FISH, immunohistochemistry, or other tests; the development of biopsy-proven extramedullary disease (e.g., CSF, testicle, lymph node, skin); or CNS relapse, defined as a CSF sample with more than 5 WBCs per high-power field with lymphoblasts on cytospin, or two consecutive CSF specimens meeting the CNS-2 criteria (<5 WBC/µL with lymphoblasts) obtained at least three weeks apart. Participants alive without disease relapse are censored at date of last disease evaluation (which can include clinical evaluation and blood counts, does not require a bone marrow examination).
Median Disease-Free Survival (DFS) | Up to 10 years
  DFS based on Kaplan-Meier method is defined as the time from confirmed complete remission (CR) to the earlier of relapse or death due to any cause. Relapse is defined as the presence of more than 5% lymphoblasts in bone marrow confirmed by flow cytometry, cytogenetics, FISH, immunohistochemistry, or other tests; the development of biopsy-proven extramedullary disease (e.g., CSF, testicle, lymph node, skin); or CNS relapse, defined as a CSF sample with more than 5 WBCs per high-power field with lymphoblasts on cytospin, or two consecutive CSF specimens meeting the CNS-2 criteria (<5 WBC/µL with lymphoblasts) obtained at least three weeks apart. Participants who are alive without disease relapse are censored at the date of last disease evaluation.
Median Overall Survival (OS) | Up to 10 years
  Overall Survival (OS) based on Kaplan-Meier method is defined as the time from registration to death due to any cause or censored at date last known alive.
Rate of Allogeneic Transplantation | CR can be documented either at the end of Induction IA (32 days) or Induction IB (74 days).
  Rate of allogeneic transplantation is defined as the proportion of participants who undergo allogeneic transplantation while in their first complete remission (CR).
Reason of Allogeneic Transplantation | CR can be documented either at the end of Induction IA (32 days) or Induction IB (74 days).
  This outcome measures the number of participants who undergo allogeneic transplantation in their first complete remission (CR) and the reasons for transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Marlise R Luskin, MD, MSCE, Principal Investigator — Dana-Farber Cancer Institute

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu